CLINICAL TRIAL: NCT01420107
Title: Video Recording in the Delivery Room in Very Preterm Infants (Video Apgar Trial)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Helmut Küster, MD, University Children's Hospital, Greifswald
Other Study IDs: 123456789
Record Dates: First submitted 2011-02-16; First posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Premature Birth
Keywords: Infant, Premature; Delivery Rooms; Video Recording; Outcome Assessment (Health Care)
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A video of the delivery room management will be taken using standardized conditions. The video will be evaluated either locally by those directly involved in the delivery room care of this specific infant or anonymously at the main study center. Using a standardized evaluation form a set of predefined interventions is rated regarding at what time they took place and at what time they should have taken place. The difference in time for all interventions is summed up to a score. This score should allow to assess the delivery room management in comparison to the desired standard as well as between hospitals. The evaluation forms of all centers will be analyzed at the main study center to define correlations between certain delivery room interventions and short term outcome.

Aim of the study is to

* gather data on how delivery room care is currently done,
* come closer to an agreement between different NICUs towards what should be done in the delivery room under what circumstances in which way,
* find those interventions with potential influence on short term outcome. Those aspects of management that are different between centers and show correlation with short term outcome will be the focus of future prospective intervention trials in order to find the best way how to take care of preterm infants in the delivery room.

Hypothesis:

In preterm infants <32;0 weeks of gestational age a correlation exists between specific delivery room interventions and short term outcome.

DETAILED DESCRIPTION:
Delivery room interventions measured are: Stimulation, Ventilation, Oxygen, Cardiac massage, Suctioning, ven / art access, fluid and drugs given

Short term outcome measurements are: IVH, PVL, Pneumothorax, BPD, DOL when first time 120mL/kg oral feeds, NEC, ROP, death, Head circumference at discharge

ELIGIBILITY:
Inclusion Criteria:

* preterm infants <32;0 weeks of gestational age

Exclusion Criteria:

* Infants in whom no life support is being planned - e.g. those with lethal malformations

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm infants <32;0 weeks of gestational age
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The Delivery Room Management Score (DRMS) negatively correlates with short term outcome (none of (death, IVH °3 or 4, PVL, pneumothorax, BPD, NEC °2 or 3, ROP °3 to 5)) | Outcome is measured at first discharge from your hospital
  On special request by the PRS-Team: this is any time between 1 Minute of life in case of delivery room death and up to 2 and more years in case of several complications during the hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Küster, MD, Principal Investigator — University Children's Hospital of Greifswald, Germany
Locations (1):
- University Children's Hospital, Greifswald, Germany